CLINICAL TRIAL: NCT02661971
Title: Perioperative RAMucirumab in Combination With FLOT Versus FLOT Alone for reSEctable eSophagogastric Adenocarcinoma - RAMSES - a Phase II/III Trial of the AIO
Brief Title: FLOT vs. FLOT/Ramucirumab for Perioperative Therapy of Gastric or GEJ Cancer (RAMSES)
Acronym: RAMSES/FLOT7
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Institut für Klinische Krebsforschung IKF GmbH at Krankenhaus Nordwest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RAMSES/FLOT7
Record Dates: First submitted 2016-01-19; First posted 2016-01-25 (Estimated); Last update posted 2022-07-11 (Actual); Status verified 2022-07

CONDITIONS: Stomach Cancer; Gastroesophageal Junction Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Docetaxel; Oxaliplatin; Leucovorin; Fluorouracil; Ramucirumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FLOT alone (Active Comparator): Pre-operative therapy with FLOT followed by surgical resection followed by post-operative therapy with FLOT
  * Docetaxel 50 mg/m², d1
  * Oxaliplatin 85 mg/m², d1
  * Calciumfolinat 200 mg/m², d1
  * 5-Fluorouracil 2600 mg/m², d1
  Interventions: Drug: Docetaxel; Drug: Oxaliplatin; Drug: Calciumfolinat; Drug: 5-Fluorouracil
- FLOT + Ramucirumab (Experimental): Pre-operative therapy with FLOT + ramucirumab followed by surgical resection followed by post-operative therapy with FLOT + ramucirumab
  * Ramucirumab 8mg/kg, d1
  * Docetaxel 50 mg/m², d1
  * Oxaliplatin 85 mg/m², d1
  * Calciumfolinat 200 mg/m², d1
  * 5-Fluorouracil 2600 mg/m², d1
  Interventions: Drug: Docetaxel; Drug: Oxaliplatin; Drug: Calciumfolinat; Drug: 5-Fluorouracil; Biological: Ramucirumab

INTERVENTIONS:
Drug: Docetaxel — Docetaxel 50 mg/m², d1
  Other Names: TAXOTERE®
Drug: Oxaliplatin — Oxaliplatin 85 mg/m², d1
  Other Names: ELOXATIN®
Drug: Calciumfolinat — Leucovorin 200 mg/m², d1
  Other Names: Leucovorin
Drug: 5-Fluorouracil — 5-FU 2600 mg/m², d1
  Other Names: 5-FU
Biological: Ramucirumab — Ramucirumab 8mg/kg, d1
  Arms: FLOT + Ramucirumab

SUMMARY:
Previous studies provide a strong theoretical rationale for the conduct of a randomized study evaluating the efficacy and safety of ramucirumab in combination with FLOT in the perioperative treatment of resectable adenocarcinoma of the stomach or GEJ.

DETAILED DESCRIPTION:
This is a multicenter, randomized, controlled, open-label study including patients with locally advanced adenocarcinoma of the stomach and GEJ scheduled to receive perioperative chemotherapy.

The scope of the phase II portion of the trial is to evaluate pathological response rates of either regimen assessed by a centralized pathology and evaluate safety and tolerability.

Patients with locally advanced esophagogastric adenocarcinoma (i.e. cT2 any N or any T N-positive) with exclusion of distant metastases will be included in this trial.

Patients will be centrally reviewed and then stratified by tumor site (GEJ vs. gastric), histological type (intestinal vs. diffuse/mixed or unknown) and clinical stage (T1/2 vs. T3/4 and/or N+) and randomized 1:1 to receive either FLOT (Arm A) or FLOT/ramucirumab (Arm B).

Arm A (FLOT) Patients randomized to Arm A will receive 4 pre-operative cycles (8 weeks) of biweekly FLOT (Docetaxel 50 mg/m² in 250 ml NaCl 0.9%, iv over 1 h; Oxaliplatin 85 mg/m² in 500 ml G5%, iv over 2h; Leucovorin 200 mg/m² in 250 ml NaCl 0.9%, iv over 30 min; 5-FU 2600 mg/m², iv over 24 h, q2wk) of the preoperative treatment phase. Surgery in Arm A is planned to occur 4 to 6 weeks after d1 of last FLOT. Patients will receive 4 additional post-operative cycles (8 weeks) of FLOT in the post-operative treatment phase. Post-operative treatment should start 6 to 8 weeks, but at maximum 12 weeks after surgery.

Arm B (FLOT/ramucirumab) Patients randomized to Arm B will receive ramucirumab 8mg/kg i.v. over 60 min in combination with the FLOT regimen, which is administered identical to Arm A as described above. Surgery in Arm B is planned to occur 4 to 6 weeks after d1 of last FLOT/ramucirumab dose (but never earlier than 4 weeks after d1 of last FLOT/ramucirumab dose). Patients will receive 4 additional post-operative cycles (8 weeks) of FLOT/ramucirumab in the post-operative treatment phase followed by a total of 16 cycles of ramucirumab as a monotherapy (q2wk), starting 2 weeks after d1 of the last cycle of FLOT/ramucirumab.

In both of the arms, tumor assessments (CT or MRI) are performed before randomization and prior to surgery, and then every 3 months thereafter until progression/relapse, death or end of follow-up. A change from CT into MRI in the follow up period is possible at any time.

During treatment, clinical visits (blood cell counts, detection of toxicity) occur prior to every treatment dose. Safety of FLOT/ramucirumab will be monitored continuously by careful monitoring of all adverse events (AEs) and serious adverse events (SAEs) reported.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed, resectable adenocarcinoma of the gastroesophageal junction (AEG/GEJ-type II-III) or the stomach (uT2, uT3, uT4, any N category, M0), or any T N+ M0 patient, with the following specifications:

   1. Medical and technical operability, according to the techniques described in Chapter 12 Surgical Therapy that are subtotal, total or transhiatal extended gastrectomy (patients planned to receive transthoracic esophagectomy are not eligible for the study)
   2. Participating sites in PETRARCA study: Negative HER-2 detection (score IHC HER-2 0 or IHC HER-2 1+ ); IHC HER-2 2+ and negative by FISH, SISH or CISH1
2. No preceding cytotoxic or targeted therapy
3. No prior partial or complete tumor resection
4. Female and male patients ≥ 18 and ≤ 70 years. Patients in reproductive age must be willing to use adequate contraception during the study and for 7 months after the end of ramucirumab treatment (Appropriate contraception is defined as surgical sterilization (e.g., bilateral tubal ligation, vasectomy), hormonal contraception (implantable, patch, oral), and double-barrier methods (any double combination of: IUD, male or female condom with spermicidal gel, diaphragm, sponge, cervical cap)). Female patients with childbearing potential need to have a negative pregnancy test within 7 days before study start.
5. ECOG ≤ 1
6. Exclusion of distant metastasis by CT or MRI of abdomen, pelvis, and thorax, bone scan or MRI (if bone metastases are suspected due to clinical signs). Exclusion of the infiltration of any adjacent organs or structures by CT or MRI.
7. Laparoscopic exclusion of peritoneal carcinomatosis, in case of ascites, peritoneal masses, or if otherwise suspected clinically
8. Adequate hematological, hepatic and renal function parameters:

   1. Leukocytes ≥ 3000/mm³, platelets ≥ 100,000/mm³, neutrophil count (ANC) ≥1000/µL, hemoglobin ≥9 g/dL (5.58 mmol/L),
   2. Adequate coagulation function as defined by International Normalized Ratio (INR) ≤ 1.5, and a partial thromboplastin time (PTT) ≤ 5 seconds above the ULN (unless receiving anticoagulation therapy). Patients receiving warfarin/phenprocoumon must be switched to low molecular weight heparin and have achieved stable coagulation profile prior to randomization.
   3. Serum creatinine ≤ 1.5 x upper limit of normal
   4. Urinary protein ≤1+ on dipstick or routine urinalysis (UA; if urine dipstick or routine analysis is ≥2+, a 24-hour urine collection for protein must demonstrate <1000 mg of protein in 24 hours to allow participation in this protocol).
   5. Bilirubin ≤ 1.5 x upper limit of normal, AST and ALT ≤ 3.0 x upper limit of normal, alkaline phosphatase ≤ 6 x upper limit of normal
9. Patient able and willing to provide written informed consent and to comply with the study protocol and with the planned surgical procedures

Exclusion Criteria:

1. Known hypersensitivity against ramucirumab, 5-FU, leucovorin, oxaliplatin, or docetaxel
2. Other known contraindications against ramucirumab, 5-FU, leucovorin, oxaliplatin, or docetaxel
3. Patients with esophageal cancer and those with adenocarcinoma of GEJ type I and all patients who are planned to have transthoracic esophagectomy.
4. Clinically significant active coronary heart disease, cardiomyopathy or congestive heart failure, peripheral artery occlusive disease (PAOD, German pAVK), or any history of aortic aneurysm
5. Any arterial thromboembolic events, including but not limited to myocardial infarction, transient ischemic attack, cerebrovascular accident, or unstable angina.
6. Uncontrolled or poorly-controlled hypertension (>160 mmHg systolic or > 100 mmHg diastolic for >4 weeks) despite standard medical management.
7. Clinically significant valvular defect
8. Past or current history of other malignancies not curatively treated and without evidence of disease for more than 5 years, except for curatively treated basal cell carcinoma of the skin and in situ carcinoma of the cervix
9. Criteria of unresectability, e.g.:

   * Radiologically documented evidence of major blood vessel invasion or encasement by cancer.
   * Patients with involved retroperitoneal (e.g. para-aortal, paracaval or interaortocaval lymph nodes) or mesenterial lymph nodes (distant metastases!)
10. Known brain metastases
11. Other severe internal disease or acute infection
12. Peripheral polyneuropathy ≥ NCI Grade II
13. Chronic inflammatory bowel disease
14. Grade 3-4 GI bleeding within 3 months prior to enrollment.
15. History of gastric perforation or fistulae in past 6 months
16. Serious or nonhealing wound, ulcer, or bone fracture within 28 days prior to enrollment.
17. The patient has undergone major surgery within 28 days prior to enrollment except staging laparoscopy.
18. Receiving chronic antiplatelet therapy, including aspirin (Once-daily aspirin use (maximum dose 325 mg/day) is permitted), nonsteroidal anti-inflammatory drugs (including ibuprofen, naproxen, and others), dipyridamole or clopidogrel, or similar agents.
19. History of deep vein thrombosis, pulmonary embolism, or any other significant thromboembolism (venous port or catheter thrombosis or superficial venous thrombosis are not considered "significant") during the 3 months prior to randomization.
20. Cirrhosis at a level of Child-Pugh B (or worse) or cirrhosis (any degree) and a history of hepatic encephalopathy or ascites.
21. On-treatment participation in another clinical study in the period 30 days prior to inclusion and during the study
22. Subject pregnant or breast feeding, or planning to become pregnant within 7 months after the end of treatment.
23. Patients in a closed institution according to an authority or court decision (AMG § 40, Abs. 1 No. 4)
24. Any other concurrent antineoplastic treatment including irradiation
25. Current chronic alcohol, nicotine or drug abuse or history of chronic alcohol abuse during last 12 months. Nicotine abuse is defined as ≥ 25 pack-years (Willigendael et al., 2004).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2021-12 (Actual); Study Completion 2022-06-20 (Actual)

PRIMARY OUTCOMES:
Phase II: Rate of pathological complete or subtotal responses (pCR/pSR): assessed according to Becker remission criteria | 3 years
Phase III: Overall Survival (OS): time from randomization to death of any cause | 3 years
  Survival rates for the different time points will be determined using the Kaplan-Meier analysis of OS.

SECONDARY OUTCOMES:
Phase II/III: R0 resection rate: reported descriptively | 75 days
Phase II/III: Progression Free Survival (PFS): time from randomization until disease progression, disease recurrence after surgery or death of any cause | 3 years
  Survival rates for the different time points will be determined using the Kaplan-Meier analysis of PFS
Phase II: Overall Survival (OS): time from randomization to death of any cause | 3 years
Phase III: Pathological response rates: assessed according to Becker remission criteria (Becker et al., 2003) | 75 days
Phase III: Progression Free Survival (PFS): time from randomization until disease progression, disease recurrence after surgery or death of any cause | 3/5 years
Phase III: Overall Survival (OS): time from randomization to death of any cause | 3/5 years
Phase II/III: Subgroup analyses: pCR/pSR according to subgroup (intestinal vs. diffuse/mixed or unknown and GEJ vs. gastric) | 3/5 years
Phase II/III: Subgroup analyses: OS (medians and rates) according to subgroup (intestinal vs. diffuse/mixed or unknown and GEJ vs. gastric) | 3/5 years
Phase II/III: Subgroup analyses: PFS (medians and rates) according to subgroup (intestinal vs. diffuse/mixed or unknown and GEJ vs. gastric) | 3/5 years

CONTACTS AND LOCATIONS:
Overall Officials: Salah-Eddin Al-Batran, Prof. Dr., Principal Investigator — Institute of Clinical Cancer Research (IKF), UCT - University Cancer Center
Locations (2):
- Institute for Clinical Cancer Research Krankenhaus Nordwest, Frankfurt, Germany
- Università degli studi della Campania "Luigi Vanvitelli", Napoli, Campania, Italy

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared.

REFERENCES:
- [Derived] Goetze TO, Hofheinz RD, Gaiser T, Schmalenberg H, Strumberg D, Goekkurt E, Angermeier S, Zander T, Kopp HG, Pink D, Siegler G, Schenk M, de Vita F, Galizia G, Maiello E, Bechstein WO, Elshafei M, Loose M, Sookthai D, Brulin T, Pauligk C, Homann N, Al-Batran SE. Perioperative FLOT plus ramucirumab for resectable esophagogastric adenocarcinoma: A randomized phase II/III trial of the German AIO and Italian GOIM. Int J Cancer. 2023 Jul 1;153(1):153-163. doi: 10.1002/ijc.34495. Epub 2023 Mar 23. PMID 36883420